CLINICAL TRIAL: NCT04836065
Title: European Society Of Intensive Care Medicine COVID-19 Project (UNITE-COVID)
Brief Title: ESICM UNITE COVID-19 Project (UNITE-COVID)
Acronym: UNITE-COVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ESICMUNITE2020
Record Dates: First submitted 2020-06-25; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: COVID-19 Infection
Keywords: Covid-19; Infection; Inflammation; respiratory distress; coagulation; thromboembolus; rehabilitation; renal; cardiac; mobilization
MeSH Terms: conditions — COVID-19; Infections; Inflammation; Dyspnea; Thrombosis; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is arguably the biggest challenge critical care medicine has been confronted with since its conception. Critical care services around the world are flooded by patients presenting with severe respiratory failure who require prolonged treatment in the ICU. Despite the support provided, outcomes are poor, particularly in ventilated patients.

Many unanswered questions remain regarding the pathophysiology of COVID-19, particularly in severely ill patients. No evidence-based treatment is currently available, yet different often experimental therapies are administered to patients.

As experience grows, new phenotypes are recognized, and unreported complications are observed in the most severely ill patients. Although many registries are currently including patients, few of them focus on ICU patients and their specific treatments and newly observed complications and challenges.

Although the pandemic may appear on its return in many countries that are now easing the restrictions that were put in place to limit the spread of the disease, it can be expected that COVID-19 will be a continued challenge in ICUs globally until a safe and effective vaccine is found. Efforts to study the disease should continue in order to advance our understanding of the disease as well as improve treatment options.

DETAILED DESCRIPTION:
This is a multicenter, international, anonymized point prevalence study. Patients who were present in the ICU on the day in April 2020 with the highest number of COVID-19 patients in the unit. Data can be entered in the database until July 2020. Retrospective data collection and entry is allowed.

Subjects believed to fulfill all eligibility criteria, and none of the exclusion criteria, detailed in the relevant section of this protocol, will be included in the study.

Data will be entered in the database anonymously.

Data will consist of two core elements:

1. Center data (to be completed once)
2. Patient data

For different domains with specific, highly relevant and un(der)explored ICU research questions, an focused data set is to be completed. These domains include:

1. Respiratory
2. Coagulation and thrombo-embolic events
3. Infectious complications
4. Rehabilitation
5. Renal

ELIGIBILITY:
Inclusion Criteria:

* Patient is present in an ICU or in any other place of the hospital under the care of the critical care team on the day between 15th February 2020 and 15th June 2020 with the highest number of COVID-19 patients in the unit. The exact date can be decided by the local investigator.
* COVID-19 confirmed diagnosis through PCR or equivalent diagnostic technique

Exclusion Criteria:

* Any of the following is regarded as a criterion for exclusion from the study: SARS-CoV2 positive without COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19 infection present in the ICUs of participating hospitals or in any other place of the hospital under the care of the critical care team on the day between 15th February 2020 and 15th June 2020 with the highest number of COVID-19 patients in the unit or in any other place of the hospital under the care of the critical care team (date to be decided by local investigator).
Sampling Method: Probability Sample
Enrollment: 4995 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients admitted with confirmed COVID19 infection | One day with 60 day follow-up
  Number of patients in the ICU on the study day
Mortality (ICU) | One day with 60 day follow-up
  Proportion of patients who have died at ICU discharge
Mortality (60-day) | One day with 60 day follow-up
  Proportion of patients who have died at day 60

SECONDARY OUTCOMES:
Duration of hospitalization in the ICU | One day with 60 day follow-up
  Length of stay in the ICU
Proportion of patients requiring invasive mechanical ventilation | One day with 60 day follow-up
  Proportion of patients who require invasive mechanical ventilation during ICU stay versus all patients
Proportion of patients developing infections during ICU stay | One day with 60 day follow-up
  Proportion of patients who acquire an infection during their ICU stay versus all patients
Proportion of patients developing thromboembolic events during ICU stay | One day with 60 day follow-up
  Proportion of patients who develop any thromboembolic event during their ICU stay versus all patients
Proportion of patients requiring tracheotomy during ICU stay | One day with 60 day follow-up
  Proportion of patients who are require a tracheostomy versus all patients

CONTACTS AND LOCATIONS:
Overall Officials: Jan DE WAELE, Principal Investigator — University of Gent Hospital
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lodigiani C, Iapichino G, Carenzo L, Cecconi M, Ferrazzi P, Sebastian T, Kucher N, Studt JD, Sacco C, Bertuzzi A, Sandri MT, Barco S; Humanitas COVID-19 Task Force. Venous and arterial thromboembolic complications in COVID-19 patients admitted to an academic hospital in Milan, Italy. Thromb Res. 2020 Jul;191:9-14. doi: 10.1016/j.thromres.2020.04.024. Epub 2020 Apr 23. PMID 32353746
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Derived] Kloss P, Lindholz M, Milnik A, Azoulay E, Cecconi M, Citerio G, De Corte T, Duska F, Galarza L, Greco M, Girbes ARJ, Kesecioglu J, Mellinghoff J, Ostermann M, Pellegrini M, Teboul JL, De Waele J, Wong A, Schaller SJ; ESICM UNITE COVID Investigators. Early mobilisation in critically ill COVID-19 patients: a subanalysis of the ESICM-initiated UNITE-COVID observational study. Ann Intensive Care. 2023 Nov 14;13(1):112. doi: 10.1186/s13613-023-01201-1. PMID 37962748
- [Derived] Conway Morris A, Kohler K, De Corte T, Ercole A, De Grooth HJ, Elbers PWG, Povoa P, Morais R, Koulenti D, Jog S, Nielsen N, Jubb A, Cecconi M, De Waele J; ESICM UNITE COVID investigators. Co-infection and ICU-acquired infection in COIVD-19 ICU patients: a secondary analysis of the UNITE-COVID data set. Crit Care. 2022 Aug 3;26(1):236. doi: 10.1186/s13054-022-04108-8. PMID 35922860